CLINICAL TRIAL: NCT04889742
Title: Hyperthermia Enhanced Re-irradiation of Loco-regional Recurrent Tumors
Acronym: HETERERO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Sebastian Zschaeck, MD, PI, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HETERERO
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Recurrent Cancer; Prostate Cancer; Cervical Cancer; Anal Cancer; Sarcoma; Rectal Cancer; Neuroendocrine Tumors; Esophageal Cancer; Pancreas Cancer; Squamous Cell Carcinoma
Keywords: re-irradiation; hyperthermia; local recurrence; hyperthermic
MeSH Terms: conditions — Recurrence; Prostatic Neoplasms; Uterine Cervical Neoplasms; Anus Neoplasms; Sarcoma; Rectal Neoplasms; Neuroendocrine Tumors; Esophageal Neoplasms; Pancreatic Neoplasms; Carcinoma, Squamous Cell; Hyperthermia; Fever

STUDY DESIGN:
Intervention Model Description: Patients will receive additional hyperthermia according to physicians´choice as a radiosensitizer to standard of care re-irradiation or re-chemoradiation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Hyperthermia (Experimental): Patients will receive 6-8 treatments additional loco-regional hyperthermia concurrent to re-irradiation. Hyperthermia will start on the third day of fractionated radiotherapy and will be given twice per week. According to site of recurrent disease either deep-regional, capacitive or superficial hyperthermia devices may be used.
  Interventions: Device: loco-regional hyperthermia

INTERVENTIONS:
Device: loco-regional hyperthermia — loco-regional hyperthermia by the use of microwave, capacitive, or superficial hyperthermia devices.

SUMMARY:
This study investiagates deep-regional or superficial hyperthermia to enhance radiotherapy or chemoradiation in patients that suffer recurrent disease after previous radiotherapy.

DETAILED DESCRIPTION:
patients that present a relapse within the previously irradiated volume can be included in this trial. These patients will receive re-irradiation according to clinical guidelines and hyperthermia as study intervention. According to tumor location hyperthermia can either be performed by microwave or by capacitive devices.

The primary endpoint of this study is non-inferiority of re-irradiation compared to the initial course of radiotherapy (calculated as time to local failure).

ELIGIBILITY:
Inclusion Criteria:

* prior radiotherapy of the treatment side with a treatment dose > 30 Gray (Gy) EQD2 (calculated with alpha/beta value of 9)
* local/ regional / or oligometastatic tumor recurrence. Maximum number of three macroscopic tumor lesions with at least one of them receiving prior radiotherapy
* macroscopic tumor recurrence
* side of recurrence is amenable to hyperthermia (abdomen, pelvis, extremities, spine, cervical lymphnodes)
* planned re-irradiation dose of at least 40 Gy EQD2 (calculated with alpha/beta value of 9)

Exclusion Criteria:

* >3 macroscopic tumor lesion
* brain metastases
* recurrence is amenable to local ablative radiotherapy (brachytherapy or stereotactic radiotherapy)
* recurrence region is not amenable to hyperthermia (lung, liver, mediastinum)
* contraindications for hyperthermia (serious cariovascular disease, ICD or larger implants at the treatment site)
* psychiatric disorders that impede proper informed consent
* serious comorbidities with very limited prognosis quo ad vitam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-05-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Local tumor recurrence | 3 years
  Local tumor recurrence of re-irradiated lesions, calculated with the Kaplan-Meier estimates. Local recurrence after hyperthermic re-irradiation will be compared to time-to recurrence after initial treatment.

SECONDARY OUTCOMES:
Overall survival | 3 years
  Overall survival after start of re-irradiation
Progression-free survival | 3 years
  Progression-free survival after start of re-irradiation
Freedom from distant metastases | 3 years
  Freedom from distant metastases after start of re-irradiation
Patient reported quality of Life | 3 years
  patient reported quality of life measured by the EORTC qlq-c30 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Zschaeck, MD, Principal Investigator — Charité
Locations (1):
- Klinik für Radioonkologie und Strahlentherapie, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No